CLINICAL TRIAL: NCT01022346
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Multicenter Study of the Safety and Response Rate of 3 Subcutaneously Administered Doses of 5 X 10^7 PFU RO5217790 in Patients With High Grade Cervical Intraepithelial Neoplasia Grade 2 or 3 Associated With High Risk HPV Infection
Brief Title: A Study of RO5217790 in Participants With High Grade Cervical Intraepithelial Neoplasia (CIN) Associated With High Risk Human Papillomavirus (HR-HPV) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV25025; 2008-006946-24 (EudraCT Number)
Record Dates: First submitted 2009-11-20; First posted 2009-12-01 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Cervical intraepithelial neoplasia; RO5217790
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Placebo matched to RO5217790 will be administered subcutaneously on Days 1, 8, and 15.
  Interventions: Drug: Placebo
- RO5217790 (Experimental): RO5217790 will be administered at a dose of 5*10^7 plaque forming unit (pfu) subcutaneously on Days 1, 8, and 15.
  Interventions: Drug: RO5217790

INTERVENTIONS:
Drug: Placebo — Placebo matched to RO5217790 will be administered subcutaneously on Days 1, 8, and 15.
  Arms: Placebo
Drug: RO5217790 — RO5217790 will be administered at a dose of 5*10^7 pfu subcutaneously on Days 1, 8, and 15.
  Arms: RO5217790

SUMMARY:
This randomized, double-blind, placebo-controlled, parallel arm study will assess the safety and the efficacy of RO5217790 on histologic resolution in participants with high grade CIN associated with HR-HPV infection. Participants will be randomized to receive 3 subcutaneous injections of either placebo or RO5217790 on Days 1, 8, and 15. Study assessments will be made at Baseline, at Month 3 and 6, and every 6 months thereafter for an overall of 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis within 2 months prior to the first dose of RO5217790 of CIN 2/3 confirmed by colposcopy-directed punch biopsy; patients must have at least 1 quadrant of residual CIN2/3 disease remaining after biopsy. Entry to the trial will be allowed based on the local assessment of this criterion; however, CIN 2/3 diagnosis will have to be confirmed by the central pathologist for the purposes of analyzing the study
* Have satisfactory colposcopy, i.e. the entire acetowhite or disease area as well as the entire squamocolumnar junction visualized by colposcopy
* Have detection at screening of a single or multiple HR-HPV infection by analysis of liquid based cytology (LBC) material on the Roche Linear Array assay consistent with any of the trial strata as specified in study protocol

Exclusion Criteria:

* Have colposcopically visible CIN2/3 disease extending over more than 2 quadrants
* Have any anatomical condition of the cervix, including that resulting from previous cervical surgery, congenital malformation or other condition, that would interfere with a complete evaluation of the transformation zone and surveillance of CIN. If an endocervical curettage (ECC) is performed, and the endocervical curettings reveal CIN, patients are eligible as long as the endocervical lesion is directly extending from the primary lesion and is colposcopically visible in its entirety
* Have vulvar (VIN) or vaginal (VAIN) intraepithelial neoplasia
* Have atypical endometrial or glandular cells or evidence of carcinoma on biopsy
* Have a serious, concomitant disorder, including active systemic infection requiring treatment
* Have a prior history of or current malignancy other than adequately treated skin cancer (squamous cell cancer or basal cell carcinoma), unless the history of skin cancer is at the site of study treatment administration
* Have a proven or suspected immunosuppressive disorder or autoimmune disease
* Have any significant cardiac, hepatic or renal disease
* Have active viral infections including human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis B virus (HBV), cytomegalovirus (CMV), and Epstein barr virus (EBV) within 30 days of receiving study treatment. Mild viral infections such as Herpes Simplex Virus 1 (HSV-1) or common cold are not excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2009-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with CIN2/CIN3 associated with HPV16 single infection who achieved Histologic resolution (Defined as no CIN), determined by evaluation of tissue derived from surgical excision | Month 6

SECONDARY OUTCOMES:
Percentage of participants who achieved Histologic resolution (Defined as no CIN), determined by evaluation of tissue derived from surgical excision | Months 6
Percentage of participants who achieved Histologic response (Defined as CIN Grade less than [<] 2), determined by evaluation of tissue derived from surgical excision | Month 6
Percentage of participants with viral clearance based on Roche Linear assay results | Months 3 and 6
Percentage of participants with immunologic response to HPV antigens | Day 1 (predose), Days 8, 15, and 29, Months 3 and 6
Percentage of Participants with at least one Adverse Events (AEs) | Up to Month 30

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (60):
- United States (40):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Colton, California
  - Los Angeles, California
  - Colorado Springs, Colorado
  - Stamford, Connecticut
  - Washington D.C., District of Columbia
  - Lake Worth, Florida
  - Miami, Florida
  - Plantation, Florida
  - Sarasota, Florida
  - South Miami, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Decatur, Georgia
  - Marrero, Louisiana
  - Framingham, Massachusetts
  - Kansas City, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Lawrenceville, New Jersey
  - Brightwaters, New York
  - The Bronx, New York
  - New Bern, North Carolina
  - Winston-Salem, North Carolina
  - Englewood, Ohio
  - Gallipolis, Ohio
  - Oklahoma City, Oklahoma
  - West Reading, Pennsylvania
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Myrtle Beach, South Carolina
  - Nashville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - McAllen, Texas
  - Sandy City, Utah
  - Norfolk, Virginia
- Belgium (6):
  - Antwerp
  - Brussels
  - Edegem
  - Ghent
  - Leuven
  - Tienen
- Finland (4):
  - Hus
  - Kuopio
  - Oulu
  - Tampere
- France (6):
  - Bordeaux
  - Dijon
  - Nantes
  - Paris
  - Reims
  - Strasbourg
- San Juan, Puerto Rico
- Spain (3):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Bilbao, Vizcaya